CLINICAL TRIAL: NCT03543358
Title: A Multicenter, Long-Term, Rollover Extension Study of Rovalpituzumab Tesirine
Brief Title: A Long-Term Study of Rovalpituzumab Tesirine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-291
Expanded Access: NCT03503890 (No longer available)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: rovalpituzumab tesirine; rollover study; cancer
MeSH Terms: conditions — Neoplasms | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Post-Treatment Follow-Up/Optional Retreatment (Experimental): Arm A includes participants who enter the extension study while in post-treatment follow-up. This arm includes optional rovalpituzumab tesirine retreatment plus dexamethasone per participant per retreatment period.
  Interventions: Drug: rovalpituzumab tesirine
- Arm B: Continued Treatment (Experimental): Arm B includes participants who enter the extension study while receiving ongoing rovalpituzumab tesirine treatment plus dexamethasone in the parent study.
  Interventions: Drug: rovalpituzumab tesirine

INTERVENTIONS:
Drug: rovalpituzumab tesirine — Optional retreatment with rovalpituzumab tesirine (0.3 mg/kg or previously adjusted dose) administered intravenously once every 6 weeks beginning on Day 1 (day of dosing) for 2 dose cycles
  Other Names: SC16LD6.5
  Arms: Arm A: Post-Treatment Follow-Up/Optional Retreatment
Drug: rovalpituzumab tesirine — Rovalpituzumab tesirine (0.3 mg/kg or previously adjusted dose) administered intravenously once every 6 weeks beginning on Day 1 (day of dosing). Subjects will receive rovalpituzumab tesirine on Day 1 of each 6-week cycle, omitting every third cycle until disease progression or study drug discontinuation.
  Other Names: SC16LD6.5
  Arms: Arm B: Continued Treatment

SUMMARY:
The purpose of this long-term, extension study is to provide ongoing safety and efficacy follow-up of subjects who participated in a rovalpituzumab tesirine study that has completed the primary analysis and that is closing.

ELIGIBILITY:
Inclusion Criteria:

* Subject had enrolled, participated in, and received at least 1 dose of rovalpituzumab tesirine in a parent study.
* Additional eligibility criterion for Arm A: subjects who discontinued the study drug in the parent study have completed the treatment emergent adverse event reporting window.

For subjects who elect optional retreatment in Arm A, must meet additional criteria before receiving rovalpituzumab tesirine retreatment including:

* Tolerated their initial 2 doses of rovalpituzumab tesirine.
* Achieved clinical benefit as defined by stable disease or better, and is determined that the subject would potentially benefit from additional treatment.
* Experienced radiographic disease progression at least 12 weeks after the second dose of rovalpituzumab tesirine.
* Received no other systemic anti-cancer therapy after rovalpituzumab tesirine treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, kidney, and liver function, per protocol.
* In subjects with central nervous system (CNS) metastases, documentation of stable or improved status as described in the protocol.

Exclusion Criteria:

* Subjects not previously enrolled in a rovalpituzumab tesirine study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (3):
- United States (3):
  - Arizona Oncology Associates, PC-HOPE (Rudasill) /ID# 204818, Tucson, Arizona
  - City of Hope National Medical Center /ID# 204885, Duarte, California
  - Univ of Pittsburgh Med Ctr /ID# 204763, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This rollover follow-up extension study was conducted in 3 sites in the United States. Participants enrolled while in post-treatment follow-up in parent studies SCRX001-002 (NCT02674568) and SCRX001-007 (NCT02874664).
Groups:
- Arm A: Post-Treatment Follow-Up/Optional Retreatment: Participants who entered the extension study while in post-treatment follow-up of parent study. Participants may receive optional retreatment with rovalpituzumab tesirine (0.3 mg/kg or previously adjusted dose) administered intravenously once every 6 weeks beginning on Day 1 (day of dosing) for 2 dose cycles (retreatment may be repeated).
- Arm B: Continued Treatment: Participants who entered the extension study while receiving ongoing rovalpituzumab tesirine treatment plus dexamethasone in the parent study. Participants receive rovalpituzumab tesirine (0.3 mg/kg or previously adjusted dose) on Day 1 of each 6-week cycle, omitting every third cycle until disease progression or study drug discontinuation.
Period: Overall Study
Arm/Group | Arm A: Post-Treatment Follow-Up/Optional Retreatment | Arm B: Continued Treatment
Started | 3 | 0
Received Treatment or Retreatment | 0 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Parent Study Closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Arm A: Post-Treatment Follow-Up/Optional Retreatment
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Treatment or Retreatment Who Experience a Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either a reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. TEAEs and serious TEAEs are defined as any event that began or worsened in severity after the first dose of study drug. For more details on AEs, please see the Adverse Event section.
Time Frame: From first dose of study drug until 70 days following last dose of study drug; up to approximately 5 years.
Population: No participants received treatment or retreatment in this study.
Arm/Group | Arm A: Post-Treatment Follow-Up/Optional Retreatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 13.6 months (maximum time on study)
Arm/Group | Arm A: Post-Treatment Follow-Up/Optional Retreatment
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Post-Treatment Follow-Up/Optional Retreatment (N=3)
Insomnia (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03543358/Prot_SAP_000.pdf